CLINICAL TRIAL: NCT02553980
Title: Development and Dissemination of an Online Exercise and Health Promotion Program for Hong Kong Middle-aged Chinese: The Virtual Trainer System 3rd Version
Brief Title: Virtual Trainer System (3rd Version) for Physical Activity Promotion in Middle-aged Hong Kong Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Stanley Sai-Chuen Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KPF14ICF14
Record Dates: First submitted 2015-02-17; First posted 2015-09-18 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Sedentary Lifestyle
Keywords: Physical activity; Information technology; Middle-aged; Health promotion
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: From 1,300 recruitment questionnaires, 261 met inclusion criteria, and 119 were randomly assigned into either n=53 in group 1 (VT3 intervention), 38 in group 2 (VT2 intervention), or 28 control (no-VT).
Who Masked: Participant
Masking Description: randomly assigned into either treatment 1, treatment 2, or control. All participants were managed in individual basis, hence no interaction between any participants was guaranteed. Participants were informed only their treatment without knowing the existence of other treatment.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical activity promotion I (Experimental): Participants in this group attended the "VT3" program (with Automatic HR detection)
  Interventions: Behavioral: Follow Your Virtual Trainer (FYVT) program
- Physical activity promotion II (Experimental): Participants in this group attended the "VT2" program (self PA report)
  Interventions: Behavioral: Follow Your Virtual Trainer (FYVT) program
- Control (Placebo Comparator): Participants in this group did not receive any VT treatment, and live as usual.
  Interventions: Other: Daily PA recommendation & healthy lifestyle suggestions

INTERVENTIONS:
Behavioral: Follow Your Virtual Trainer (FYVT) program — Participants in intervention group will under the instruction of a web-based computer software termed "Virtual Trainer", which interact with their smartphone apps, to conduct a 3-month self-planned PA training program. A serious of online video seminars related to healthy lifestyle advice will be released to the participants among 3 months. After that, 6 months observation will be followed.
  Arms: Physical activity promotion I; Physical activity promotion II
Other: Daily PA recommendation & healthy lifestyle suggestions — A written advice of daily PA recommendation, and the textual content of the healthy lifestyle seminars will be provided to the participants.
  Arms: Control

SUMMARY:
Practicing a habitual physical activity is important for health. A Virtual Trainer (VT) online system was developed in 2006 (1st version) and improved in 2010 (2nd version) for encouraging an active lifestyle. This project intends to further improve the VT (3rd version) which incorporates more effective psychological and e-health theories, and disseminate it to Hong Kong middle-aged adults.

DETAILED DESCRIPTION:
Hong Kong is a highly urbanized city that many people work long hours daily and over the week, especially for those middle-aged adults. The limited time and lack of professional exercise instruction are always the barriers for them to participate in physical activity (PA). With the advances in information technology (IT), the knowledge of PA can be rapidly disseminated through the Internet and smartphone. We design an IT- instruction based lifestyle intervention program, with the purpose to improve PA level and health status in a sample of middle-aged Hong Kong adults. A two-arm parallel individual level randomized controlled trial (RCT) named "Follow Your Virtual Trainer (FYVT)" will be conducted among 200 healthy and sedentary Chinese adults aged from 40 to 65 years. The participants will be randomly allocated into intervention group or control group. Those in intervention group will under the instruction of a web-based computer software termed "Virtual Trainer", which interact with their smartphone apps, to conduct a 3-month self-planned PA training program. A serious of online video seminars with healthy lifestyle themes will be released to the participants biweekly among 3 months. After that, 6 months observation will be followed. Those in control group will only receive a written advice of standard PA recommendation, and the textual content of the seminars. The assessments will be implemented at baseline, 3, 6, and 9 month. Primary outcome is PA measured by accelerometer and International Physical Activity Questionnaire; the second outcomes include cardio-respiratory fitness, resting energy expenditure, anthropometrics, body composition, blood pressure, health-related quality of life, sleep quality and quantity, fatigue, behavior mediators, and maintenance of PA.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 to 65 years
* able to understand Cantonese and read Chinese
* self-reported inactivity (no habitual exercise experience for at least 6 months)
* the baseline resting energy expenditure (REE) is less than 1.05 kcal•min-1 for men and 0.85 kcal•min-1 for women
* reachable by telephone
* have basic computer skills
* have smartphone and always surf internet (at least 4 times per week)
* will not leave Hong Kong for a long time (longer than 2 months) during the study period

Exclusion Criteria:

* self-reported history of cardiovascular and pulmonary diseases, neurological disorder, musculo-skeletal disorder, and osteoarthritis
* receiving medically prescribed diet or PA intervention
* blood pressure ≥ 160/100 mmHg
* using of medication that may influence exercise performance
* for women, currently pregnant or plan to become pregnant in the next 1 years, and those receiving hormonal therapy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Changes of physical activity level as measures by accelerometer and International Physical Activity Questionnaire | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months

SECONDARY OUTCOMES:
Changes of cardio-respiratory fitness as measured by the symptom limited maximal treadmill exercise test using the metabolic analyzer (Cosmed K4b2, Italy) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
  The maximal oxygen intake (VO2 max in ml•min-1•kg-1) is used as indicator of cardio-respiratory fitness in our study.
Changes of resting VO2 (ml•min-1•kg-1) as measured by the metabolic analyzer (Cosmed K4b2, Italy) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of resting kilocalorie expenditure (KCal in KCal•min-1) as measured by the metabolic analyzer (Cosmed K4b2, Italy) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of resting heart rate (HR in beats•min-1) as measured by heart rate monitor | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of body weight as measured by weighting scale | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of body mass index (BMI) as measured by the calculation of weight (kg) divided by the square of height (cm) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of waist circumference as measured by standardized tape measure | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of hip circumference as measured by standardized tape measure | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of body fat percentage as measured by the bioelectrical impedance analysis (Tanita, BC 581, Japan) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of body mass as measured by the bioelectrical impedance analysis (Tanita, BC 581, Japan) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of waist hip ratio (WHR) as measured by the calculation of dividing the waist circumference (cm) by the hip circumference (cm) | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of blood pressure as measured by the mercury sphygmomanometer | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of health-related quality of life as measured by the SF-36 | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of sleep quality as measured by the Pittsburgh Sleep Quality Index | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of sleep quantity as measured by a 7-day Daily Sleep Log | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Changes of self-perceived fatigue as measured by the Numeric Rating Scale (NRS)-fatigue | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
Maintenance of physical activity as measured a self-administered questionnaire | Measures will be done at two time points: 6 months and 9 months
  A self-administered questionnaire will be given to the participants at 3 and 6 months to evaluate their maintenance of physical activity.
Behavior mediators as measured by a self-administered questionnaire | Measures will be done at four time points: baseline, 3 months, 6 months, and 9 months
  The possible behavior mediators will be examined by a self-administered questionnaire that bases on Ajzen's guideline for developing a Theory of Planned Behavior questionnaire. We will structure these mediator variables according to attitude, subjective norms and perceived behavioral control, to understand their intention to active participation in physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Sai-chuen Hui, EdD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Hui SS, Xie YJ, Kwok RC, Tam EW, Mak WWS, Mo PK. Follow Your Virtual Trainer (FYVT): a randomised controlled trial protocol of IT-based lifestyle intervention programme to promote physical activity and health among middle-aged Hong Kong Chinese. BMJ Open. 2018 Feb 3;8(2):e017908. doi: 10.1136/bmjopen-2017-017908. PMID 29431125